CLINICAL TRIAL: NCT03131908
Title: Phase I/II Study of the Selective PI3K-Beta Inhibitor GSK2636771 in Combination With Pembrolizumab in Patients With Metastatic Melanoma and PTEN Loss
Brief Title: Study of the Selective PI3K-Beta Inhibitor GSK2636771 in Combination With Pembrolizumab in Patients With Metastatic Melanoma and PTEN Loss
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH); Merck Sharp & Dohme LLC (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0774; NCI-2018-01609 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Melanoma and Other Malignant Neoplasms of Skin; Metastatic Melanoma
Keywords: Melanoma and other malignant neoplasms of skin; Metastatic Melanoma; GSK2633771; Pembrolizumab; Keytruda; MK-3475; SCH-900475
MeSH Terms: conditions — Melanoma | interventions — GSK2636771; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GSK2636771 + Pembrolizumab (Experimental): Phase I: Participants receive the lowest dose level of GSK2636771. Each new group receives a higher dose of GSK2636771 than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of GSK2636771 is found. Participants receive the same dose level of Pembrolizumab.
  Phase II: Participants receive GSK2636771 at the highest dose that was tolerated in Phase 1. Participants receive the same dose level of Pembrolizumab.
  Interventions: Drug: GSK2636771; Drug: Pembrolizumab

INTERVENTIONS:
Drug: GSK2636771 — Phase I Starting Dose of GSK2636771: 300 mg by mouth given for 21 days.
  Phase II Dose of GSK2636771: Maximum tolerated dose from Phase I.
Drug: Pembrolizumab — Phase I and II Dose of Pembrolizumab: 200 mg given by vein every 3 weeks.
  Other Names: Keytruda; MK-3475; SCH-900475

SUMMARY:
The goal of this clinical research study is to learn if GSK2636771 given in combination with pembrolizumab can help to control the disease in patients with refractory (has not responded to treatment) metastatic melanoma. The safety of this drug combination will also be studied.

This is an investigational study. Pembrolizumab is FDA approved and commercially available and FDA approved for the treatment of several types of cancer, including melanoma. GSK2636771 is not FDA approved or commercially available. It is currently being used for research purposes only. The study doctor can explain how the study drugs are designed to work.

Up to 41 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 3 groups of 3-6 participants will be enrolled in Phase 1 of the study, and up to 35 participants will be enrolled in Phase 2.

If you have metastatic cancer, you may be enrolled in Phase 1 of this study. If you have metastatic melanoma, you may be enrolled in Phase 1 or Phase 2 of this study.

If you are enrolled in Phase 1, the dose of GSK2636771 in combination with pembrolizumab you receive will depend on when you join this study. The first group of participants will receive the lowest dose level of GSK2636771. Each new group will receive a higher dose of GSK2636771 than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of GSK2636771 is found.

If you are enrolled in Phase 2, you will receive GSK2636771 at the highest dose that was tolerated in Phase 1.

All participants will receive the same dose level of pembrolizumab.

Study Drug Administration:

Every study cycle is 21 days.

* You will take GSK2636771 by mouth every day for 21 days.
* You will receive pembrolizumab by vein for 30 minutes one (1) time on Day 1 of every cycle.

You should receive the study drugs at least 1 hour before or 2 hours after eating.

Length of Study:

You may receive the study drugs for up to 2 years. If the doctor thinks it is in your best interest, you may continue to receive either GSK2636771 or pembrolizumab for 1 more year. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the Follow-Up Visits.

Study Visits:

On Day 1 of Cycles 1, 3, 5, and 7:

* You will have a physical exam.
* You will have an EKG. If the doctor thinks it is needed, you will also have an ECHO and MUGA scan.
* Blood (about 3 teaspoons) and urine will be collected for routine tests.
* Blood (about 2 tablespoons) will be drawn for pharmacokinetic (PK) testing before the dose, at 30 minutes, 1, 2, 3, 4, 6, and 24 hours after the dose. (Cycle 1 only). PK testing measures the amount of study drug in the body at different time points.
* Blood (about 2 tablespoons) will be drawn for immune function testing (Cycles 3 & 5 only).
* You will have a PET/CT scan or MRI to check the status of the disease (Cycle 5 only and then every 12 weeks after that).
* If you can become pregnant, blood (about ½ teaspoon) or urine will be collected for a pregnancy test.

On Day 1 of Cycles 2, 4, 6, 8 and beyond:

* You will have a physical exam.
* Blood (about 1½ teaspoon) and urine will be collected for routine tests.
* Blood (about 1 teaspoon) will be drawn for PK testing before the dose. (Cycle 2 only)
* If the doctor thinks it is needed, you will have an ECHO and MUGA scan.
* If you can become pregnant, blood (about ½ teaspoon) or urine will be collected for a pregnancy test.

On Day 1 of Cycles 2, 3, and 5, and every 12 weeks after that, you will be asked to have a core biopsy. Only 1 of these will be required, and the others will be optional. Though it is preferred that this be performed at Cycle 2, you and your doctor will choose which of these biopsies will be the required one.

Every 12 weeks after Cycle 5, blood (about 2½ tablespoons) will be drawn for immune system testing.

End of Study Dosing Visit:

After you stop receiving the study drugs:

* You will have a physical exam.
* If the doctor thinks it is needed, you will have an ECHO and MUGA scan.
* Blood (about 1 teaspoon) and urine will be collected for routine tests.
* If the disease got worse while you are on study, you may have a core biopsy.
* If you can become pregnant, blood (about ½ teaspoon) or urine will be collected for a pregnancy test.

Follow-Up Period:

Up to 30 days after the End-of-Study Dosing Visit and every 6 weeks:

* You will have a physical exam.
* Blood (about 2 tablespoons) and urine will be collected for routine tests.
* If the doctor thinks it is needed, you will have an ECHO and MUGA scan.
* If you can become pregnant, blood (about ½ teaspoon) or urine will be collected for a pregnancy test.

One (1) time every 12 weeks:

* You will have a PET/CT) scan or MRI to check the status of the disease.
* You will be called by a member of the study staff to check your health. These calls should last about 5 minutes each time.

Treatment Beyond Progression:

If the disease appears to be getting worse or the tumors appear to be getting larger, you may still be able to receive the study drug if you and your doctor decide it is in your best interest. Sometimes the disease appears to get worse but the study drug is actually working.

However, there are risks of continuing to receive the study drug because the disease may actually be getting worse. You are still at risk for side effects due to the study drug. This could also delay starting other treatments. The disease may get worse to the point that you are no longer able to receive other treatments.

If you choose to receive the study drug after the disease gets worse, you will continue to have study visits. The study doctor will discuss this option with you.

Alcohol and Activity Restriction:

On days when you have multiple PK blood draws, you should not have alcohol for at least 24 hours before your dose of study drug.

You should not exercise for 48 hours before each PK and/or routine testing blood draw.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Be >/= 18 years of age on day of signing informed consent.
3. Evidence of PTEN loss in tumors by IHC or molecular analysis.
4. Have measurable disease based on RECIST 1.1.
5. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
6. Patients who have unresectable Stage III through stage IV metastatic cancer who have not achieved complete or partial response after 6 months of therapy or who have progressed on PD-L1 or PD-1 directed therapy including combinations. The Phase II portion eligibility will be restricted to patients with metastatic melanoma.
7. In Phase I, Patients are allowed to have more than three prior systemic therapeutic regimens. Patients enrolled to Phase II, can have no more than three prior systemic therapeutic regimen for unresectable stage III or stage IV metastatic cancer. This includes chemotherapy, biologic therapy, biochemotherapy, or investigational treatment. This does not include any therapies given in the adjuvant setting.
8. Have a life expectancy of at least 12 weeks.
9. Have not received any chemotherapeutic, biological, investigational agent, radiation therapy, or used an investigational device within 28 days of study drug administration.
10. Able to swallow and retain orally administered medication.
11. On the dose expansion and Phase II portions of the study, patients must be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion before and at least one time point while on therapy. Correlative biopsies will be optional in the Phase I portion of the study. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1 without intervening systemic therapy.
12. Within 10 days of treatment initiation, the subject must demonstrate adequate organ function defined as follows: Absolute neutrophil count must be >/= 1500 per microliter (uL). Platelets must be >/=100,000 per uL. Hemoglobin must be >/= 9 grams per deciliter or >/= 5.6 millimoles per liter without transfusion or EPO dependency within 7 days of assessment. Serum creatinine must be </= 1.0 times the upper limit of normal (ULN) OR measured or calculated creatinine clearance per institutional standard (Glomerular Filtration Rate (GFR) can also be used in place of creatinine or CrCl) must be >/= 60 milliliters per minute OR proteinuria by urine dipstick must be </= 1+. Aspartate aminotransferase (AST) AND alanine aminotransferase (ALT) must be </= 2.5 times the ULN OR each must be </= 5 times the ULN for subjects with liver metastases. Alkaline phosphatase (ALP) must be </= 2 times the ULN. Serum
13. Cont#12 total bilirubin must be </= 2.0 milligrams per deciliter except in patients with Gilbert's disease. Direct bilirubin must be </= the upper limit of normal for subjects with total bilirubin levels > 1.5 times the upper limit of normal. Albumin must be >/= 2.5 grams per deciliter. Left ventricular ejection fraction (LVEF) must be >/= 50% by echocardiogram (ECHO) or Multigated Acquisition (MUGA) scan. International Normalized Ratio (INR) must be </= 1.5 times the upper limit of normal unless the subject is receiving anticoagulant therapy as long as prothrombin time(PT) or partial thromboplastin time(PTT) is within therapeutic range of intended use of anticoagulants.Activated partial thromboplastin time(aPTT) must be </= 1.5 times the upper limit of normal unless the subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants. Serum phosphate must be within normal limit. Serum calcium must be within normal limit
14. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
15. Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 4 months after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
16. Male subjects with a female partner of childbearing potential must agree to use acceptable methods of contraception from the time of Screening until 3 months after the last dose of study treatments.

Exclusion Criteria:

1. Patients are excluded if they have a history of or active autoimmune disease, as follows: Patients with a history of inflammatory bowel disease are excluded from this study as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]). Patients with motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome and Myasthenia Gravis) are excluded. Patients with a history of autoimmune thyroiditis are eligible if their current thyroid disorder is treated and stable with replacement or other medical therapy.
2. Has active infections or serious general medical conditions (such as active myocardial infarction (MI), cerebrovascular accident (CVA), or respiratory failure).
3. Any unresolved > Grade 1 toxicity (per CTCAE 4.0) from previous anti-cancer therapy or previously administered agent at the time of enrollment, except for alopecia, Grade 2 anemia (if hemoglobin is >9 grams per deciliter (g/dL)) Note: If the subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
4. Presence of any clinically significant gastrointestinal (GI) abnormality or other condition(s) that may alter absorption such as malabsorption syndrome or major resection of the stomach or substantial portion of the small intestine.
5. Active peptic ulcer disease or history of abdominal fistula, GI perforation, or intra abdominal abscess within 28 days prior to enrollment
6. Previous major surgery within 28 days prior to enrollment.
7. Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal or cardiac disease).
8. Has a QTc >450 milliseconds (msec) or QTc >480 msec for subjects with bundle branch block (BBB) NOTES: The QTc is the QT interval corrected for heart rate by Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machine-read or manually over-read. The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial. For purposes of data analysis QTcF will be used.
9. History or evidence of cardiovascular risk including any of the following: - Clinically significant electrocardiogram (ECG) abnormalities including second degree (Type II) or third degree atrioventricular block - History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, stenting, or bypass grafting within the past 6 months prior to enrollment - Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system - Left ventricular ejection fraction (LVEF) below 50% - Known cardiac metastases.
10. Poorly controlled hypertension (defined as systolic blood pressure [SBP] of >/= 150 millimeters of mercury (mmHg) or diastolic blood pressure [DBP] of >100 mmHg based on a mean of three measurements at approximately 2-minute intervals) NOTE: Initiation or adjustment of antihypertensive medication(s) is permitted if done thirty or more days prior to enrollment.
11. History of congenital platelet function defect (e.g., Bernard-Soulier syndrome, Chediak-Higashi syndrome, Glanzmann thrombasthenia, storage pool defect)
12. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. NOTE: Replacement dose steroids (equivalent to 10 mg prednisone) are allowed.
13. Has a known history of active TB (Bacillus Tuberculosis).
14. Hypersensitivity to Pembrolizumab or GSK2636771 or excipients.
15. Has a known prior or additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
16. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least two weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
17. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
19. Has known psychiatric or substance abuse disorders that in the opinion of the registering physician or PI would interfere with cooperation with the requirements of the trial.
20. Has a known history or positive test for Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies). Testing at the time of Screening is not required.
21. Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at time of Screening or any history of hepatitis.
22. Has received a live vaccine within 30 days of planned start of study therapy.
23. Current use of or anticipated requirement during the study of any prohibited medication(s). Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum-Tolerated Dose (MTD) of GSK2636771 in Combination with Pembrolizumab in Participants with Metastatic Melanoma and PTEN Loss | 3 weeks
  Maximum-tolerated dose defined as the highest dose where ≤ 1 out of 6 participants experiences dose limiting toxicities (DLTs).
Objective Response Rate (ORR) of GSK2636771 in Combination with Pembrolizumab in Participants with Metastatic Melanoma and PTEN Loss | 12 weeks
  Objective Response Rate (ORR) determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 in metastatic melanoma.

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
  Overall survival (OS) defined from treatment start date to date of death for any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Hussein Tawbi, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org